CLINICAL TRIAL: NCT04188613
Title: Use of High-Frequency Jet Ventilation During Percutaneous Tracheostomy as an Alternative to a Classic Mechanical Ventilation by Endotracheal Tube
Brief Title: Use of High-Frequency Jet Ventilation During Percutaneous Tracheostomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Diskapi Yildirim Beyazit Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Savas Altinsoy, Principal Investigator, Diskapi Yildirim Beyazit Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: HFJV
Record Dates: First submitted 2019-12-04; First posted 2019-12-06 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2021-01

CONDITIONS: Tracheostomy Complication; High-frequency Jet Ventilation; Percutaneous Tracheostomy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HFJV (Experimental): In preparation for the percutaneous tracheotomy, the patient was covered in a sterile fashion. The patient was extubated, and the jet ventilator catheter was inserted to trachea and ventilation will be start.
  Interventions: Device: Percutaneous tracheostomy
- ETT (Active Comparator): In preparation for the percutaneous tracheotomy, the patient was covered in a sterile fashion. Endotracheal tube (ETT) was removed through the vocal cords.
  Interventions: Device: Percutaneous tracheostomy
- LMA (Active Comparator): In preparation for the percutaneous tracheotomy, the patient was covered in a sterile fashion. Endotracheal tube (ETT) was removed and laryngeal mask airway device inserted.
  Interventions: Device: Percutaneous tracheostomy

INTERVENTIONS:
Device: Percutaneous tracheostomy — Age, gender, height, BMI, ASA scores, presence and type of additional diseases, tracheostomy day, pre- and post-procedure blood gas analysis, duration of procedure, duration of anesthesia, complications during the procedure (bleeding , desaturation, accidental extubation, malposition, bradycardia, hypotension, etc.) will be recorded from intensive care follow-up. Patients will be observed for mortality in the first 30 days after the procedure. Mortality results will be recorded.

SUMMARY:
Percutaneous tracheostomy is the mouth opening of the tracheal ostium to the skin by creating an opening in the anterior wall of the trachea using Seldinger methods. This procedure is done using an endotracheal tube (ETT) or a laryngeal mask (LMA). High-frequency jet ventilation (HFJV) commonly used in oropharyngeal surgeries and creates an extra passage for the procedure. The investigators aimed to demonstrate the effective use of HFJV in percutaneous tracheostomy.

DETAILED DESCRIPTION:
Seventy five patients between 18-80 years of age who were hospitalized in intensive care unit were included in the study. The number of patients will be finalized by power analysis. whose written consent cannot be obtained and who undergo surgical tracheostomy for any reason will be excluded from the study. In addition, patients with active infection in the area of the procedure, bleeding diathesis and pathologies that interfere with the procedure in the ultrasonographic evaluation (thyroid diseases, etc.) will be excluded from the study. Patients will be divided into three groups as those using classical ventilation (group 1), HFJV (group 2) and classical laryngeal mask (group 3). Age, gender, height, BMI, ASA scores, presence and type of additional diseases, tracheostomy day, pre- and post-procedure blood gas analysis, duration of procedure, duration of anesthesia, complications during the procedure (bleeding , desaturation, accidental extubation, malposition, bradycardia, hypotension, etc.) will be recorded. Patients will be observed for mortality in the first 30 days after the procedure. Mortality results will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* percutaneous tracheostomy procedure

Exclusion Criteria:

* whose written consent cannot be obtained
* who undergo surgical tracheostomy for any reason
* patients with active infection in the area of the procedure,
* bleeding diathesis
* pathologies that interfere with the procedure in the ultrasonographic evaluation (thyroid diseases, etc.)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
percutaneous tracheostomy time | during procedure
  the time the needle enters the skin to the insertion of the tracheostomy cannula

SECONDARY OUTCOMES:
complications rate | during procedure
  the complications such as ET cuff puncture, Difficult insertion of tracheostomy tube, Accidental extubation, Bleeding vs. during percutaneous tracheostomy

CONTACTS AND LOCATIONS:
Locations (1):
- Ministry of Health Diskapi Yıldırım Beyazıt Training and Research Hospital Ankara, Turkey, Ankara, Turkey (Türkiye)